CLINICAL TRIAL: NCT07082309
Title: The Effect of Ketone Monoesters on Skeletal Muscle Protein Synthesis and Whole-body Protein Metabolism.
Acronym: WAKM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 9482953
Record Dates: First submitted 2025-07-03; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants
Keywords: ketone monoesters; muscle protein synthesis; amino acid metabolism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Placebo with bitter agent (Bitrex), to flavour match to ketone condition, whey protein (0.3 g/kg), and milk fat (to match the caloric content of the ketone condition).
  Interventions: Dietary Supplement: Control
- Ketone monoester (Experimental): Ketone monoester ((R)-3-hydroxybutyl (R)-3-hydroxybutyrate) and whey protein (0.3 g/kg)
  Interventions: Dietary Supplement: Ketone Monoester (KE) and whey protein beverage

INTERVENTIONS:
Dietary Supplement: Ketone Monoester (KE) and whey protein beverage — Ketone monoester ((R)-3-hydroxybutyl (R)-3-hydroxybutyrate) and whey protein (0.3 g/kg)
  Arms: Ketone monoester
Dietary Supplement: Control — Placebo with bitter agent (Bitrex), to flavour match to ketone condition, whey protein (0.3 g/kg), and milk fat (to match the caloric content of the ketone condition).
  Arms: Control

SUMMARY:
The ketone β-hydroxybutyrate (BHB) is endogenously produced during periods of low glucose availability, serving as an alternative metabolic fuel. Beyond its role as an energy substrate, BHB acts as a pleiotropic signalling molecule, modulating various physiological processes across multiple tissues. BHB can also be ingested orally as a ketone monoester, transiently elevating plasma concentrations of BHB to a level similar to those seen following several days of fasting, thereby obviating the need for dietary manipulation. The influence of BHB on human skeletal muscle protein metabolism remains poorly understood, although emerging evidence suggests that BHB may play a role in regulating muscle protein turnover. As such, BHB supplementation may support skeletal muscle remodelling and offer therapeutic benefits, and investigating this is of considerable interest. This study will investigate the ability of oral BHB ingestion - co-ingested with protein - to stimulate skeletal muscle anabolism in young healthy adults. A dual amino acid stable isotope tracer approach will be utilised to determine postprandial (i.e., fed state) muscle protein synthesis (MPS) rates and whole-body amino acid kinetics, given BHBs systemic effects. This research will advance our understanding of the fundamental biology of exogenous ketosis and provide insight into the potential of BHB supplementation as a novel nutritional strategy to optimise muscle mass and quality.

DETAILED DESCRIPTION:
The ketone body β-hydroxybutyrate (BHB) is produced endogenously during periods of low glucose availability (e.g., fasting or starvation) and provides an alternative metabolic fuel. BHB also acts as a metabolic signalling molecule, modulating physiological processes across multiple tissues, including skeletal muscle. However, the impact of exogenous ketosis on muscle protein turnover, which regulates muscle mass and modulates physical function, remains largely unexplored. As such, understanding how BHB affects skeletal muscle protein turnover is fundamentally important. The ingestion of 0.5g/kg body mass BHB appreciably increases plasma BHB concentrations for several hours, to ~3-5 mM; equivalent to several days of fasting. This offers a model to exogenously elevate plasma BHB concentrations and investigate how BHB interacts with feeding to affect postprandial protein metabolism, the period primarily responsible for driving changes in muscle quality and quantity.

An early study demonstrated that the infusion of BHB stimulates muscle protein synthesis rates (MPS), whilst only a single recent study has investigated the effect of oral BHB ingestion (exogenous ketosis) on MPS. Prior work demonstrated that the ingestion of an oral ketone monoester stimulated MPS, and it did so to a similar extent as 10 g whey protein or co-ingestion of the two, in healthy young males. While this study provides useful insights, several unanswered questions/objectives that justify the need for further investigation remain:

* To determine how BHB ingestion influences myofibrillar protein synthesis, plasma amino acid concentrations, and amino acid kinetics following the co-ingestion of a physiologically relevant meal-like protein dose.
* To examine how BHB ingestion affects plasma amino acid concentrations and kinetics following protein co-ingestion, addressing prior research limitations where differences in carbohydrate intake and postprandial insulin levels confounded the independent effects of ketones.
* To assess the impact of BHB ingestion on whole-body protein metabolism following protein co-ingestion, as previous studies have not examined its potential influence on protein breakdown, amino acid kinetics, and net protein balance.
* To investigate whether BHB ingestion influences mitochondrial muscle protein synthesis following protein co-ingestion, given its established effects on mitochondrial metabolism, yet unexamined role in mitochondrial protein turnover.

The aim, therefore, is to establish the effect of BHB and protein co-ingestion on myofibrillar protein synthesis rates, mitochondrial protein synthesis rates, and whole-body protein turnover. We will address this question by utilising a meal-like bolus of protein (0.3 g/kg whey protein), with and without 0.5g/kg body mass BHB (matching the test drinks caloric content via the addition of fat to minimally stimulate insulin secretion), whilst applying a dual-stable isotope tracer approach.

ELIGIBILITY:
Inclusion Criteria:

• BMI 18-30

Exclusion Criteria:

* Body mass index (BMI) < 18.5 or > 30 kg/m2
* Age < 18 or > 40
* Regularly smokes
* Type 2 diabetes
* Cardiovascular disease, metabolic disease and hypertension (≥ 140/90 mmHg)
* Gastrointestinal disorders
* Use medicines that may impact protein metabolism or that are anti-inflammatory (determined at the screening)
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle protein synthesis rates (FSR) | 5 hours (2 hours postabsorptive, 3 hours postprandial)
  Skeletal muscle protein synthesis rates

SECONDARY OUTCOMES:
Plasma amino acid concentrations | 5 hours
  Plasma amino acid concentrations
Whole-body phenylalanine kinetics assessed by stable isotope tracer methodology, including rate of appearance (Ra), rate of disappearance (Rd), hydroxylation rate, and net balance. | 5 hours (2 hours postabsorptive, 3 hours postprandial)
  Whole-body kinetics of phenylalanine will be quantified using a primed continuous intravenous infusion of stable isotope-labelled phenylalanine and tyrosine tracers (e.g., L-[ring-²H₅]-phenylalanine and L-[³-¹³C]-tyrosine). Arterialised-venous blood samples will be collected at steady state to determine tracer enrichment in plasma.
  The following parameters will be calculated:
  Rate of appearance (Ra) of phenylalanine (μmol/kg/min), rate of disappearance (Rd) of phenylalanine (μmol/kg/min), hydroxylation rate of phenylalanine to tyrosine (μmol/kg/min) (derived from the appearance of labelled tyrosine from labelled phenylalanine), and net balance of phenylalanine (μmol/kg/min): calculated as the difference between Ra and Rd to assess overall protein balance.
Serum insulin concentrations | 5 hours
  Serum insulin concentrations
Plasma beta hydroxybutyrate concentrations | 5 hours
  Plasma beta hydroxybutyrate concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Health and Life Sciences, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No